CLINICAL TRIAL: NCT05863130
Title: A Phase I, Open-label, Two-arm, Non-randomised Trial to Investigate the Metabolism and Pharmacokinetics of a Single Dose of BI 764198 (C-14) Administered as Oral Solution Using Two Different Approaches in Healthy Male Volunteers
Brief Title: A Study in Healthy Men to Test How BI 764198 is Processed in the Body
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1434-0016
Record Dates: First submitted 2023-04-25; First posted 2023-05-17 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Healthy
MeSH Terms: interventions — Carbon-14

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BI 764198 (C-14) (approach 1) (Experimental)
  Interventions: Drug: BI 764198 (C-14) (approach 1)
- BI 764198 (C-14) (approach 2) (Experimental)
  Interventions: Drug: BI 764198 (C-14) (approach 2)

INTERVENTIONS:
Drug: BI 764198 (C-14) (approach 1) — BI 764198 (C-14) (approach 1)
  Arms: BI 764198 (C-14) (approach 1)
Drug: BI 764198 (C-14) (approach 2) — BI 764198 (C-14) (approach 2)
  Arms: BI 764198 (C-14) (approach 2)

SUMMARY:
The main objective of this trial is to investigate the basic pharmacokinetics of BI 764198 and its metabolites, total radioactivity including mass balance, excretion pathways and metabolism following oral administration to healthy male volunteers of a single oral dose of BI 764198 (C-14) in i) a classical hADME approach and ii) a hADME microtracer approach.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (Blood Pressure (BP), Pulse Rate (PR)), 12-lead ElectroCardioGram (ECG), and clinical laboratory tests
* Age of 18 to 65 years (inclusive)
* BMI of 18.5 to 29.9 kg/m2 (inclusive)
* Signed and dated written informed consent in accordance with ICH-GCP and local legislation prior to admission to the trial

Exclusion Criteria:

* Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 45 to 90 mmHg, or pulse rate outside the range of 40 to 100 bpm
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders Further exclusion criteria apply

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-05-03 (Actual); Primary Completion 2023-11-09 (Actual); Study Completion 2023-11-09 (Actual)

PRIMARY OUTCOMES:
Fraction of [14C]-radioactivity excreted in urine expressed as percentage of the administered dose over the time interval from 0 to the last quantifiable time point (feurine,0-tz) | Up to 31 days
Fraction of [14C]-radioactivity excreted in faeces expressed as percentage of the administered dose over the time interval from 0 to the last quantifiable time point (fefaeces,0-tz) | Up to 31 days

SECONDARY OUTCOMES:
Maximum measured concentration of the analyte in plasma (Cmax) | Up to 31 days
Area under the concentration-time curve of the analyte over the time interval from 0 to the last quantifiable data point) in plasma (AUC0-tz) | Up to 31 days

CONTACTS AND LOCATIONS:
Locations (1):
- ICON, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com